CLINICAL TRIAL: NCT06421467
Title: Insulin Injection Practices in People With Diabetes in Spain
Brief Title: Insulin Injection Practices in Spain
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Francisco Javier Ampudia Blasco, Principal Investigator, Fundación para la Investigación del Hospital Clínico de Valencia
Other Study IDs: EPID-ES
Record Dates: First submitted 2024-01-19; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this era of pharmaceutical and technological advancements, gaining insights into prevalent insulin administration practices under real-life conditions becomes pivotal for healthcare professionals. The investigators aim to explore insulin injection habits through an online survey among a broad, unselected group of participants with type 1 and type 2 diabetes undergoing daily prandial and/or basal insulin treatment. Eligible participants will access and complete the survey at their convenience after providing online informed consent within the study period

DETAILED DESCRIPTION:
HYPOTHESIS The study hypothesis posits that there is significant variability in the practices of insulin administration among patients with diabetes using daily insulin injections. This diversity in administration practices may have a notable impact on the overall efficacy of treatment regimens and the successful management of the disease, thereby emphasizing the need for a comprehensive understanding of these practices to enhance patient outcomes and optimize diabetes care.

OBJECTIVES The main objective of the study is to comprehensively assess and characterize the diverse insulin administration practices among individuals with diabetes using injections, focusing on both prandial and basal insulin. By employing an online survey methodology and targeting a broad demographic through a diabetes information platform Canal Diabetes, the investigators aim to gain valuable insights into the variability, challenges, and overall patterns of insulin administration. The findings will contribute to a better understanding of real-world practices, facilitating improvements in patient guidance and optimizing diabetes care strategies.

STUDY DESIGN The study follows a cross-sectional observational design, allowing the investigators to capture a snapshot of the current insulin administration practices via an online questionnaire among the diverse population of diabetes patients using multiple insulin injections.

STUDY PROCEDURE AND SCHEDULE The study, focusing on insulin administration practices among participants with diabetes using multiple insulin injections, will employ a two-month online survey accessible on the designated online platform Canal Diabetes. Recruitment efforts through the diabetes information platform Canal Diabetes will inform eligible participants about the study's voluntary nature, emphasizing response confidentiality. Participants meeting the criteria, will access and complete the online informed consent and survey at their convenience within the designated two-month period. Post-survey, collected data will be securely stored and anonymized for subsequent analysis.

STUDY DURATION The anticipated duration of this study will be 4 months, with subject recruitment set to begin in July 2024 and aiming for the completion of statistical analysis by the 31st of October 2024.

GOOD CLINICAL PRACTICE The procedures set out in this study protocol, pertaining to the conduct, evaluation, and documentation of this study, are designed to ensure that the sponsor and investigator (in this case the same person) comply with the principle of the good clinical practice guidelines and the Declaration of Helsinki in the conduct, evaluation and documentation of this study. The study will also be carried out in keeping with local legal requirements.

SUBJECTS INFORMATION AND INFORMED CONSENT Prior to taking the online questionnaire, participants will be required to provide explicit consent to participate in the study. An online informed consent document, encompassing details about the study and the consent form, will be prepared and supplied to participants. This document will be presented in a language accessible to participants, and clear contact information will be provided for any questions that may arise.

ENSURING DATA CONFIDENTIALITY The study database will not contain any information that could allow the individual identification of the study participants. The data obtained will be used exclusively for the purposes described in this research project. The information will be treated as confidential and will be stored and processed in accordance with the provisions of EU Regulation 2016/679 of the European Parliament and the Council of 27 April 2016 on the protection of personal data and the free movement of such data, as well as Organic Law 3/2018 of December.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or above
* Individuals diagnosed with diabetes (type 1 or type 2 diabetes)
* Individuals receiving multiple daily doses of insulin

Exclusion Criteria:

* Individuals utilizing continuous subcutaneous insulin infusion
* Individuals engaging in sensor-augmented pump therapy
* Individuals using automatic insulin delivery systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18 or above, diagnosed with either Type 1 or Type 2 diabetes, who actively incorporate insulin injections-both prandial and basal-into their treatment plan, with a minimum requirement of at least one injection of prandial insulin and/or basal insulin.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Number of total insulin injections | through study completion, an average of 16 weeks
  Number of total insulin injections per day
Number of prandial insulin injections | through study completion, an average of 16 weeks
  Number of prandial insulin injections per day
Number of basal insulin injections | through study completion, an average of 16 weeks
  Number of basal insulin injections per day
Timing of prandial insulin injection | through study completion, an average of 16 weeks
  Timing of prandial insulin injection: before meals, during meals, after meals, or at some point during the day
Time interval before prandial insulin injection | through study completion, an average of 16 weeks
  If insulin administration occurs before starting the meal: time interval (minutes)
Time interval after prandial insulin injection | through study completion, an average of 16 weeks
  If insulin administration occurs after the meal: time interval (minutes)
Insulin overdosing | through study completion, an average of 16 weeks
  Insulin overdosing when correcting abnormal glucose values (Y/N)
Insulin underdosing | through study completion, an average of 16 weeks
  Insulin overdosing when correcting abnormal glucose values (Y/N)
Insulin administration site | through study completion, an average of 16 weeks
  Insulin administration site: abdomen, thigh, arm
Site rotation | through study completion, an average of 16 weeks
  Injection site rotation: (Yes/No)
Change of the insulin needle | through study completion, an average of 16 weeks
  Frequency in the change of the insulin needle
Use of smart pens | through study completion, an average of 16 weeks
  Use of smart pens (Y/N)
Type of prandial insulin | through study completion, an average of 16 weeks
  Type of prandial insulin used
Daily dose of prandial insulin | through study completion, an average of 16 weeks
  Daily dose of prandial insulin (IU/kg)
Type of basal insulin | through study completion, an average of 16 weeks
  Type of basal insulin used
Daily dose of basal insulin | through study completion, an average of 16 weeks
  Daily dose of basal insulin (IU/kg)
Last HbA1c | through study completion, an average of 16 weeks
  Last HbA1c value
Date of last HbA1c | through study completion, an average of 16 weeks
  Date of last HbA1c value
Diabetic ketoacidosis | through study completion, an average of 16 weeks
  Diabetic ketoacidosis (DKA) in the last year (Y/N)
Hypoglycemic episodes | through study completion, an average of 16 weeks
  Severe hypoglycemic episodes in the last year (Y/N)
Hyperglycemic episodes | through study completion, an average of 16 weeks
  Hyperglycemic episodes with medical support in the last year (Y/N)
Age of diabetes onset | through study completion, an average of 16 weeks
  Age of diabetes onset (years/months)
Self-monitoring of capillary glucose | through study completion, an average of 16 weeks
  Self-monitoring of capillary blood glucose (SMBG) (Y/N)
Glucose monitoring in real-time or intermittently scanned | through study completion, an average of 16 weeks
  Continuous glucose monitoring (CGM) in real-time or intermittently scanned (Y/N)
Lack of daily glucose monitoring | through study completion, an average of 16 weeks
  Lack of daily glucose monitoring (Y/N)
Lack of correction based on glucose values | through study completion, an average of 16 weeks
  Lack of correction based on glucose values (Y/N)
Time in Range (%TIR) | through study completion, an average of 16 weeks
  If CGM user, CGM parameters from the last 28 days: Time in Range (%TIR)
Time Below Range (%TbR) | through study completion, an average of 16 weeks
  If CGM user, CGM parameters from the last 28 days: Time Below Range (%TbR)
Time Above Range (%TaR) | through study completion, an average of 16 weeks
  If CGM user, CGM parameters from the last 28 days: Time Above Range (%TaR)
Mean glucose (mg/dL) | through study completion, an average of 16 weeks
  If CGM user, CGM parameters from the last 28 days: mean glucose (mg/dL)
Coefficient of variation of continuous glucose sensor values (CV) | through study completion, an average of 16 weeks
  If CGM user, CGM parameters from the last 28 days: coefficient of variation of continuous glucose sensor values (CV)

CONTACTS AND LOCATIONS:
Overall Officials: F. Javier Ampudia-Blasco, Principal Investigator — HCUV-INCLIVA
Locations (1):
- INCLIVA, Valencia, Spain